CLINICAL TRIAL: NCT03241329
Title: Characterization of Normal and Pathological Oocyte Cohort After Controlled Ovarian Stimulation: Example of Endometriosis
Brief Title: Endometriosis Impact on Oocyte Quality
Acronym: EndOvo
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01163-50
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; Metabolomics; Transcriptomics; Follicular fluid; Cumulus cells; Oocyte quality
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Samples without DNA : follicular fluids
  2. Samples with DNA : cumulus cells from which RNA will be extracted in order to perform transcriptomics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case : endometriosis: Infertile patients with endometriosis that is the only cause of their infertility
- Control : tubal factor: infertile patients with tubal factor that is the only cause of their infertility

SUMMARY:
The aim of this study is to evaluate the impact of endometriosis on folliculogenesis and oocyte quality. To do so, a metabolomic approach will be conducted in order to analyze the follicular fluid. This evaluation will be completed by a transcriptomic analysis from the cumulus cells of the oocyte.

The normal and pathological oocyte cohort after controlled ovarian stimulation will be also characterized by identifying the oocyte leading to live birth.

DETAILED DESCRIPTION:
Endometriosis pathophysiology remains under controversy. Among the various issues raised, that of his involvement in an implantation failure related to an alteration of the endometrium is advanced by some authors. For others, infertility would be linked to an alteration of the oocyte quality responsible for embryonic development impairment leading to a lack of implantation. Several research groups have also mentioned the association of the two mechanisms.

The oocyte quality evaluation is also subject to controversy. Indeed, its morphological approach remains the most commonly used in routine at the IVF laboratory. However, this tool remains limited and to date, no correlation between oocyte morphology and ART outcomes have been established. In this context, there is a real need to use functional approaches such as genomics, transcriptomics, proteomics and metabolomics. However, the clinical validation and application of these functional tools have to be evaluated from a human pathology model such as endometriosis.

ELIGIBILITY:
Inclusion Criteria:

Group 1: case

a. Womens with endometriosis i. Deep endometriosis without ovarian localisation ii. Deep endometriosis associated with ovarian localisation iii. Isolated ovarian localisation b. Male partner with normal sperm parameters Group 2 : control

1. Womens with isolated tubal factor
2. Male partner with normal sperm parameters

Exclusion Criteria:

* Other pathologies responsible for female infertility
* Altered sperm parameters
* Male or female viral risk
* Oocyte or sperm donation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enrolled in a ART (assisted reproductive technology) attempt in the IVF unit of the center.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Metabolic profile | 2 years
  Identification of a possible particular metabolomic profile from the follicular fluid in endometriosis
Transcriptomic profile | 2 years
  Identification of a possible particular transcriptomic profile from the cumulus cells in endometriosis

SECONDARY OUTCOMES:
Oocyte characterization | 2 years
  Identification of a possible transcriptomic profile from the cumulus cells of the oocyte which could be predictive of live birth. Search of correlations between these profiles and (i) oocyte and embryo morphology and (ii) clinical and neonatal outcomes after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled POCATE-CHERIET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin-Port Royal, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pocate-Cheriet K, Santulli P, Kateb F, Bourdon M, Maignien C, Batteux F, Chouzenoux S, Patrat C, Wolf JP, Bertho G, Chapron C. The follicular fluid metabolome differs according to the endometriosis phenotype. Reprod Biomed Online. 2020 Dec;41(6):1023-1037. doi: 10.1016/j.rbmo.2020.09.002. Epub 2020 Sep 4. PMID 33046374